CLINICAL TRIAL: NCT01868100
Title: Preliminary Study of Financial Distress and Quality of Life in Patients With Advanced Cancer
Brief Title: Financial Distress in Patients With Advanced Cancer
Acronym: DIFIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012.762
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2013-06

CONDITIONS: Cancer; Quality of Life
Keywords: Cancer; quality of life; palliative care; supportive care; Financial distress
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- self-completion questionnaire (No Intervention)
  Interventions: Other: self-completion questionnaire

INTERVENTIONS:
Other: self-completion questionnaire

SUMMARY:
Advanced cancer has an adverse effect in virtually all dimensions of patients' lives (physical, psychosocial, spiritual, familial, role function). One of the less frequently explored effects of cancer is its impact on personal finances and the contribution of financial-related distress to overall suffering and quality of life. Financial issues have been recently found to be the second most frequent source of distress identified by cancer patients in a community cancer center context (22%).

In the context of continuous increased health care costs, it is likely that the frequency of health care related financial problems will keep rising. The relative contribution of these adverse financial events in advanced cancer patients to overall patient distress is not well assessed and this is particularly true in France. The main objective of this work is to determine the association between financial distress and quality of life of patients with advanced cancer in a Public General Hospital and in a Comprehensive Cancer Center. A secondary objective is to characterize the frequency and intensity of financial distress reported by French cancer patients and their impact on their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years old and have a diagnosis of advanced cancer which is defined as one of the following: recurrent disease, received >2 lines of chemotherapy, locally-advanced disease, metastatic disease, or refractory disease.
* Patients must have a cancer diagnosis of: breast, colon, lung or prostate.
* Patients must be able to understand, read, write, and speak French.

Exclusion Criteria:

* Clinical evidence of cognitive impairment, as determined by the palliative care physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Financial distress and quality of life | Cross sectional (one day)
  FACT-G; FACT-pal; FACT-sp for the quality of life; Self-assessment of financial distress in a 0 to 10 scale(0 no distress; 10 maximal distress)

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de soins palliatifs Groupement Hospitalier Sud, Pierre-Bénite, Pierre Bénite, France

REFERENCES:
- [Result] Barbaret C, Brosse C, Rhondali W, Ruer M, Monsarrat L, Michaud P, Schott AM, Delgado-Guay M, Bruera E, Sanchez S, Filbet M. Financial distress in patients with advanced cancer. PLoS One. 2017 May 18;12(5):e0176470. doi: 10.1371/journal.pone.0176470. eCollection 2017. PMID 28545063